CLINICAL TRIAL: NCT00140972
Title: A Multicenter, Randomized, Parallel-group, 4-Week, Double-Blind and Active Comparator-Controlled Study to Assess Efficacy, Safety, and Tolerability of Etoricoxib 60 mg Once Daily Versus Diclofenac Sodium 75 mg Twice Daily in the Treatment of Chinese Patients With Osteoarthritis of the Knee or Hip
Brief Title: A Study to Assess Etoricoxib Versus Diclofenac in Chinese Patients With Osteoarthritis of the Knee or Hip (0663-080)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-080; MK0663-080; 2005_060
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Arcoxia
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663; etoricoxib / Duration of Treatment:4 Weeks
Drug: Comparator: diclofenac sodium tablet 75 mg / Duration of Treatment:4 Weeks

SUMMARY:
A Study to Assess Etoricoxib versus Diclofenac in Chinese Patients with Osteoarthritis of the Knee or Hip

ELIGIBILITY:
Inclusion Criteria:

* Chinese males or females at least 40 years of age with osteoarthritis of the knee or hip

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-12-03 (Actual); Primary Completion 2005-06-27 (Actual); Study Completion 2005-06-27 (Actual)

PRIMARY OUTCOMES:
WOMAC pain subscale

SECONDARY OUTCOMES:
WOMAC Physical function subscale; WOMAC Stiffness subscale; Patient Global Assessment of Response to Therapy; Investigator Global Assessment of Disease Status

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Zhang F, Li Z, Yang N, Wu D, Sun L, Wu H. The clinical study of etoricoxib in the treatment of Chinese patients with osteoarthritis: a randomized double-blind trial. Chinese J of Rheum. 2013;17(5):307-312.